CLINICAL TRIAL: NCT03471637
Title: How do Self-compassion and Psychological Flexibility Mediate Change in a Compassion-Focused Therapy Group for Chronic Pain?
Brief Title: Compassion-Focused Therapy for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S0815692
Record Dates: First submitted 2017-11-06; First posted 2018-03-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain; Psychological Distress
Keywords: Chronic Pain; Compassion-Focused Therapy; Self-Compassion; Psychological Flexibility
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassion-Focused Therapy (Experimental): Compassion-Focused Therapy 11 weeks of Compassion-Focused Therapy [based on "Compassion-Focused Therapy for Dummies" (Welford, 2016)]
  Interventions: Other: Compassion-Focused Therapy

INTERVENTIONS:
Other: Compassion-Focused Therapy — Compassion-Focused Therapy 11 weeks of Compassion-Focused Therapy [based on "Compassion-Focused Therapy for Dummies" (Welford, 2016)]

SUMMARY:
This research aims to study how Compassion-Focused Therapy (CFT) might work for people with chronic pain. People with chronic pain may feel shameful about their condition and this type of therapy aims to help people to view themselves and their difficulties in a kinder, less critical way (i.e. self-compassion). Currently, no research is available on the effectiveness of CFT in helping people with chronic pain.

Participants attending a CFT-incorporated Pain Management Programme will complete a battery of questionnaires at the start of the group (week 1), in the middle of the group (week 5) and at the end of the group (week 11).

DETAILED DESCRIPTION:
Pain Management Programmes help people to manage their pain and improve quality of life, and this research will look into the processes by which this happens. This study will look at two psychological concepts: 'self-compassion' (kindness to self) and 'psychological flexibility' (willingness to tolerate difficult experiences in order to meet meaningful goals). These concepts help in understanding how people think about themselves in the context of pain.

Principle Research Question: Do self-compassion and psychological flexibility mediate change (anxiety/depression/well-being) in a Compassion-Focused Therapy group for adults with chronic pain?

Primary Outcome Measure: Strength of mediation effects

Sample Size:

[Reference 1] propose guidelines for recommended sample sizes in order to detect mediation effects with .8 power. These guidelines are informed by existing literature in the field. There is less robust research on self-compassion and chronic pain, therefore, this calculation is based on research in psychological flexibility and chronic pain.

[Reference 2] conducted correlational analyses on the processes of psychological flexibility following a group intervention based on ACT. These processes included acceptance of pain, mindfulness, psychological acceptance and values-based action (r values between 0.33 and 0.55). These positive correlations indicate that the group intervention was related to higher levels of psychological flexibility.

[Reference 3]'s review identified several studies that reported correlational effect sizes between acceptance, and depression/anxiety/daily functioning related to chronic pain (r = -0.58/-0.66/0.47 respectively). These negative correlations illustrate that higher levels of psychological flexibility were related to better outcomes.

Based on these correlational effect sizes, guidelines in [Reference 1] suggest that a sample size of 53-71 is required.

Analysis:

The analysis will focus on the proposed mediating factors (self-compassion and psychological flexibility) and how they explain the outcome of the CFT-incorporated group intervention. In order to study the processes of change, this study will measure change in mediators and outcomes over the course of the group.

In a mediation model, the effect of the independent variable (IV; CFT group) on a dependent variable (DV; outcome/change in symptoms) is conveyed through a third mediating variable. In order to be a mediator, a variable must change during the intervention, be associated with the intervention, and have an impact on the outcome.

In this study, it is hypothesised that self-compassion and/or psychological flexibility are the mediating variables that explain the influence of the group intervention on eventual outcome, i.e. the overall change in symptoms at the end of the group. Linear regression and nonparametric bias-corrected bootstrap, which corrects for skew in the data, will be applied to the data using SPSS, using the PROCESS macro. An effect of mediation will be indicated if the confidence interval does not contain zero.

Missing data will be handled using either the maximum likelihood or multiple imputation method, as recommended in literature.

ELIGIBILITY:
Please note this study is only recruiting people who have been referred and accepted onto NHS Lothian's Pain Management Programme (part of the Lothian Pain Service at the Astley Ainslie Hospital).

Inclusion Criteria:

* Fluency of English sufficient for participation in the group and completion of questionnaires
* Aged 18+ (no upper age limit)
* Ability to provide informed consent (as defined by the Five Statutory Principles of the Mental Capacity Act, Code of Practice, 2007)

Exclusion Criteria:

* Active substance misuse
* Active suicidality
* Terminal illness
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Strength of Self-Compassion as a mediator at Week 11 | Week 1
Strength of Psychological Flexibility as a mediator at Week 11 | Week 1

SECONDARY OUTCOMES:
Self-Compassion Scale (short form, SCS-SF; Neff, 2003) | [Time Frame: Week 1 (start), Week 5 (middle) and Week 11 (end) of group therapy]
  Minimum score: 12; maximum score: 60; higher score indicates higher level of self-compassion
Multi-Dimensional Psychological Flexibility Inventory (short form, MPFI-SF; Rolffs et al., 2016) | [Time Frame: Week 1 (start), Week 5 (middle) and Week 11 (end) of group therapy]
  Minimum score: 24; maximum score 144; higher score indicates higher level of psychological flexibility
The Brief Pain Inventory (short form, BPI-SF; Cleeland & Ryan, 1994) | [Time Frame: Week 1 (start), Week 5 (middle) and Week 11 (end) of group therapy]
  Minimum score: 0; maximum score 110; higher score indicates greater level of pain severity and pain interference (severity max 40 / interference max 70)
The Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) (Tennant et al., 2007) | [Time Frame: Week 1 (start), Week 5 (middle) and Week 11 (end) of group therapy]
  Minimum score: 7; maximum score: 35; higher score indicates greater level of wellbeing
The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) | [Time Frame: Week 1 (start), Week 5 (middle) and Week 11 (end) of group therapy]
  Minimum score: 0; maximum score: 42; higher score indicates higher level of anxiety and depression (anxiety max 21 / depression max 21)

CONTACTS AND LOCATIONS:
Overall Officials: Su Tin, Principal Investigator — University of Edinburgh
Locations (1):
- Astley Ainslie Hospital, Edinburgh, Edinburgh City, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fritz MS, Mackinnon DP. Required sample size to detect the mediated effect. Psychol Sci. 2007 Mar;18(3):233-9. doi: 10.1111/j.1467-9280.2007.01882.x. PMID 17444920
- [Background] McCracken LM, Gutierrez-Martinez O. Processes of change in psychological flexibility in an interdisciplinary group-based treatment for chronic pain based on Acceptance and Commitment Therapy. Behav Res Ther. 2011 Apr;49(4):267-74. doi: 10.1016/j.brat.2011.02.004. Epub 2011 Feb 15. PMID 21377652
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03471637/Prot_SAP_002.pdf
  • Informed Consent Form (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03471637/ICF_003.pdf